CLINICAL TRIAL: NCT02477735
Title: The Effect of Tympanostomy Tube Insertion on Sleep in Children With Chronic Otitis Media With Effusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-15-GF-0021-15-CTIL
Record Dates: First submitted 2015-05-21; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Otitis Media With Effusion; Sleep Disturbances
MeSH Terms: conditions — Parasomnias | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Infants with COME who will be referred for TTI will undergo actigraphy for 7 consecutive nights prior to TTI and for 7 consecutive nights 4-6 weeks following TTI.
  Interventions: Device: Actigraphy
- Healthy infants: Healthy infants that were recruited from the community well-baby clinics.

INTERVENTIONS:
Device: Actigraphy — Actigraphy will be conducted for each participant for 7 consecutive nights prior to TTI and for 7 consecutive nights 4-6 weeks following TTI.
  Groups: Study group

SUMMARY:
The purpose of this study is to investigate the prevalence of sleep disturbances in children with Chronic Otitis Media with Effusion (COME) and the effect of tympanostomy tube insertion (TTI) on sleep disturbances.

DETAILED DESCRIPTION:
Comparison of sleep disturbances will be between infants with Chronic Otitis Media with Effusion (COME) who will be referred for tympanostomy tube insertion (TTI) (study group) and healthy infants that were recruited from the community well-baby clinics (control group).

To evaluate sleep patterns, parents of the study group will complete two validated sleep questionnaires assessing the infant's typical sleep patterns based on parental reports. A week before TTI and 1 week to 1 month after the surgery, sleep will be evaluate by actigraph for a week long.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-36 months
* Referred for tympanostomy tube insertion as a treatment for COME.

Exclusion Criteria:

* Snoring and sleep disordered breathing (SDB)
* Chronic medical condition
* referred for TTI and adenoidectomy/tonsillectomy

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with COME who will be referred for TTI.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Actigraphy measurements | Up to two years

SECONDARY OUTCOMES:
OSA-18 questionnaire score | Up to two years
Brief Infant Sleep Questionnaire (BISQ) score | Up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Gad Fishman, Doctor, Principal Investigator — Dana Children's Hospital, Tel-Aviv Sourasky Medical Center, Sackler School of Medicine Tel-Aviv Univesity, Israel
Locations (1):
- "DANA" children's hospital, Tel Aviv, Israel